CLINICAL TRIAL: NCT01090323
Title: A One Year Open Label, Non-comparative Extension to a Randomized, Multicenter, Phase II Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Effects on Liver Iron Concentration (LIC) of Repeated Doses of 5-30mg/kg/Day ICL670 Relative to Deferoxamine (DFO) in Sickle Cell Disease (SCD) Patients With Transfusional Hemosideresis (THS) [Amendment 3: Extension Prolonged to 4-years]
Brief Title: Evaluation of the Safety, Tolerability, Pharmacokinetics (PK) and Effects on Liver Iron Concentration of ICL670 Relative to Deferoxamine(DFO).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0109E1; EudraCT no. 2004-000597-31 (Registry Identifier: EudraCT); NCT00171197 (obsolete NCT alias)
Record Dates: First submitted 2010-03-15; First posted 2010-03-19 (Estimated); Results first posted 2011-01-20 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-05

CONDITIONS: Sickle Cell Disease
Keywords: Deferasirox; ICL670A; Iron chelators; Sickle Cell Disease; Transfusional Hemosiderosis
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICL670 (Experimental)
  Interventions: Drug: ICL670

INTERVENTIONS:
Drug: ICL670 — Daily doses of ICL670 were taken orally 30 minutes before breakfast. The doses range from 5-40 mg/kg and were determined based on the patient's trend in serum ferritin over time during the core study (0109) and on the frequency of blood transfusions the patient received. The treatment duration was up to 4 years.

SUMMARY:
The safety, tolerability, effects on liver iron concentration and pharmacokinetics of ICL670 is studied in sickle cell disease patients with transfusional hemosiderosis.

DETAILED DESCRIPTION:
The treatment period started once the patient completed the core study and signed informed consent. It is continued for up to 4 years. Safety parameters were assessed every 4 weeks. Eye and Ear examinations were performed on a yearly basis. To further investigate the extent of iron overload, serum ferritin, iron, and transferrin were monitored every four weeks. The Program Safety Board monitored the safety of ICL670 during the study to evaluate and categorize any serious case reported in association with ICL670.

ELIGIBILITY:
Inclusion Criteria:

Patients were included who met the following criteria:

* Completion of the core [Study 0109]
* Serum ferritin greater than or equal to 500 µg/L
* Ability to comply with all study-related procedures, medications, and evaluations
* Sexually active post-menarche female patients must use double-barrier contraception, oral contraceptive plus barrier contraceptive, or must have undergone clinically documented total hysterectomy and/or oophorectomy, tubal ligation or be postmenopausal defined by amenorrhea for at least 12 months.
* Written informed consent and assent by the patient and or their parents or legal guardian.

Additional inclusion criteria for pediatric patients The definition of the term 'pediatric' for enrollment and study conduct was in accordance with local law. Parents or the legal guardians were fully informed by the investigator as to the requirements of the study. The pediatric patients themselves were informed according to their capabilities in a language and terms that they were able to understand. Written informed consent was obtained from their legal guardian on the patient's behalf in accordance with national legislation. If capable, all patients had to also personally sign their written informed consent.

Exclusion Criteria:

Patients who met the following criteria were to be excluded:

* History of non-compliance to medical regimens and patients who are considered potentially unreliable and/or not cooperative
* Serum creatinine above the age-appropriate upper limit of normal within one week prior to entry
* Patients with ALT ≥ 500 U/L within one week prior to entry
* Evidence of chelation-related cataracts or hearing loss within 4 weeks prior to baseline
* Pregnancy (as indicated by serum β-HCG pregnancy test for all female patients with the potential to become pregnant) and patients who are breastfeeding
* Patients treated with systemic investigational drug within 4 weeks prior to or with topical investigational drug within 7 days prior to the baseline visit

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2004-07; Primary Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- United States (31):
  - University of South Alabama College of Medicine, Mobile, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital & Research Center at Oakland, Oakland, California
  - University of Colorado Health Science Center, Denver, Colorado
  - Howard University Hospital, Washington D.C., District of Columbia
  - St Joseph Children's Hospital of Tampa, Tampa, Florida
  - Grady Hospital, Georgia Comprehensive Sickle Cell Center, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Tulane University Medical Center, New Orleans, Louisiana
  - LSUHSC Dept of Pediatrics, Shreveport, Louisiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - New York Methodist Hospital, Brooklyn, New York
  - New York Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Yasin, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - Santee Hematology/Oncology, Sumter, South Carolina
  - St. Jude's Children Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
- Novartis Investigative Site, Toronto, Canada
- France (2):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Paris
- Italy (4):
  - Novartis Investigative Site, Catania
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Roma
- Novartis Investigative Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- ICL670: Participants treated with ICL670 during the Core Study 0109(NCT00067080) and during the extension phase. ICL670 was administered orally once a day based on the participant's body weight.
- Crossover: Participants treated with Deferoxamine (DFO) during the Core Study 0109 (NCT00067080) and treated with ICL670 during the extension phase. ICL670 was administered orally once a day based on the participant's body weight.
Period: Overall Study
Arm/Group | ICL670 | Crossover
Started | 132 | 53
Completed | 43 | 19
Not Completed | 89 | 34
Not completed — Adverse Event | 12 | 2
Not completed — Abnormal Lab Values | 3 | 1
Not completed — Abnormal Test Procedure Results | 2 | 0
Not completed — Unsatisfactory therapeutic effect | 4 | 2
Not completed — Condition no longer requires drug | 5 | 4
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrew consent | 33 | 11
Not completed — Lost to Follow-up | 11 | 6
Not completed — Administrative problems | 6 | 4
Not completed — Death | 1 | 2
Not completed — Stopped end of core | 7 | 0
Not completed — Stopped end of extension 1# | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICL670 | Crossover | Total
Number analyzed (Participants) | 132 | 53 | 185
Age, Customized [Number; unit: participants]
  <12 years | 33 | 14 | 47
  12 - <16 years | 32 | 11 | 43
  16 - <65 years | 67 | 28 | 95
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 31 | 111
  Male | 52 | 22 | 74
Region of Enrollment [Number; unit: participants]
  France | 10 | 2 | 12
  United States | 110 | 46 | 156
  Canada | 0 | 1 | 1
  United Kingdom | 5 | 1 | 6
  Italy | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events After Start of ICL670
Description: Safety as assessed by the number of participants with adverse event or death after the start of ICL670.
Time Frame: 0 - 60 months
Population: The primary analysis was on Safety Analysis Set which comprised all participants who received at least one dose of ICL670 during the core/extension phase of the study. All participants previously treated with ICL670/DFO for 52weeks in the core study.
Measure: Number; unit: participants
Arm/Group | ICL670 | Crossover
Number analyzed (Participants) | 132 | 53
participants
  Adverse Events | 131 (10.66) | 49 (11.32)
  Deaths | 1 | 2

2. Secondary Outcome: Change in Serum Ferritin From Start of ICL670 to End of Study
Description: The main efficacy variable was change in serum ferritin in response to therapy with ICL670. Due to variability of serum ferritin, end of study was considered as the mean of at most the last 3 available observations after the start of ICL670.
Time Frame: 0 - 60 months
Population: The primary analysis was on Full Analysis Set which comprised all participants who received at least one dose of ICL670 during the core or the extension phase of the study. All participants previously treated with ICL670 or DFO for 52 weeks in the core study were eligible for enrollment.
Measure: Median (Full Range); unit: µg/L
Arm/Group | ICL670 | Crossover
Number analyzed (Participants) | 132 | 53
µg/L | -245.5 [-8701.3 to 7626.5] | -134.3 [-6124.0 to 5136.7]

ADVERSE EVENTS:
Arm/Group | ICL670 | Crossover
Serious Adverse Events (participants affected / at risk) | 97/132 | 34/53
Other Adverse Events (participants affected / at risk) | 129/132 | 47/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICL670 (N=132) | Crossover (N=53)
Acute chest syndrome (Blood and lymphatic system disorders) | 5 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 2 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypersplenism (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 | 1
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 48 | 19
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 14 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 5
Asthenia (General disorders) | 0 | 1
Catheter related complication (General disorders) | 0 | 2
Catheter site haemorrhage (General disorders) | 0 | 1
Catheter site pain (General disorders) | 1 | 1
Catheter thrombosis (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 8 | 4
Chills (General disorders) | 1 | 1
Facial pain (General disorders) | 1 | 0
Granuloma (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Necrosis (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 6 | 1
Pyrexia (General disorders) | 25 | 9
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 7 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic sequestration (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Adenovirus infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 3 | 2
Catheter bacteraemia (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 5 | 2
Cellulitis (Infections and infestations) | 3 | 1
Central line infection (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Mononucleosis syndrome (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 13 | 3
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 3 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Citrate toxicity (Injury, poisoning and procedural complications) | 1 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 0
Device failure (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 3 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Biopsy liver (Investigations) | 1 | 0
Blood alkaline phosphatase (Investigations) | 1 | 0
Blood amylase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood iron increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Pregnancy test positive (Investigations) | 1 | 0
Total lung capacity decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Complex partial seizures (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 7 | 2
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Enuresis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Breast swelling (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 3 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Catheter placement (Surgical and medical procedures) | 1 | 0
Catheter removal (Surgical and medical procedures) | 1 | 0
Central venous catheterisation (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Jugular vein distension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ICL670 (N=132) | Crossover (N=53)
Leukocytosis (Blood and lymphatic system disorders) | 4 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 8 | 2
Tachycardia (Cardiac disorders) | 2 | 3
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 37 | 13
Ear pain (Ear and labyrinth disorders) | 8 | 3
Ocular icterus (Eye disorders) | 11 | 6
Vision blurred (Eye disorders) | 9 | 5
Abdominal discomfort (Gastrointestinal disorders) | 9 | 2
Abdominal pain (Gastrointestinal disorders) | 32 | 13
Abdominal pain upper (Gastrointestinal disorders) | 27 | 15
Constipation (Gastrointestinal disorders) | 28 | 7
Diarrhoea (Gastrointestinal disorders) | 39 | 19
Dyspepsia (Gastrointestinal disorders) | 8 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 52 | 19
Toothache (Gastrointestinal disorders) | 9 | 4
Vomiting (Gastrointestinal disorders) | 45 | 17
Asthenia (General disorders) | 7 | 1
Chest pain (General disorders) | 24 | 15
Chills (General disorders) | 9 | 4
Fatigue (General disorders) | 22 | 7
Oedema peripheral (General disorders) | 14 | 4
Pain (General disorders) | 16 | 6
Pyrexia (General disorders) | 45 | 22
Jaundice (Hepatobiliary disorders) | 6 | 3
Bronchitis (Infections and infestations) | 8 | 1
Cellulitis (Infections and infestations) | 2 | 3
Ear infection (Infections and infestations) | 9 | 1
Gastroenteritis (Infections and infestations) | 12 | 3
Gastroenteritis viral (Infections and infestations) | 8 | 4
Influenza (Infections and infestations) | 14 | 4
Nasopharyngitis (Infections and infestations) | 37 | 16
Oral herpes (Infections and infestations) | 8 | 1
Pharyngitis (Infections and infestations) | 12 | 4
Pharyngitis streptococcal (Infections and infestations) | 7 | 4
Pneumonia (Infections and infestations) | 2 | 3
Rhinitis (Infections and infestations) | 9 | 0
Sinusitis (Infections and infestations) | 17 | 5
Staphylococcal infection (Infections and infestations) | 7 | 1
Tonsillitis (Infections and infestations) | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 43 | 19
Urinary tract infection (Infections and infestations) | 20 | 3
Viral infection (Infections and infestations) | 11 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 3
Excoriation (Injury, poisoning and procedural complications) | 8 | 0
Skin laceration (Injury, poisoning and procedural complications) | 4 | 3
Transfusion reaction (Injury, poisoning and procedural complications) | 8 | 2
Alanine aminotransferase increased (Investigations) | 6 | 4
Aspartate aminotransferase increased (Investigations) | 8 | 3
Blood creatinine increased (Investigations) | 12 | 4
Serum ferritin increased (Investigations) | 8 | 4
Transaminases increased (Investigations) | 9 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 3
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 8 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 48 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 41 | 13
Dizziness (Nervous system disorders) | 17 | 7
Headache (Nervous system disorders) | 61 | 30
Hypoaesthesia (Nervous system disorders) | 7 | 1
Migraine (Nervous system disorders) | 7 | 4
Anxiety (Psychiatric disorders) | 7 | 3
Depression (Psychiatric disorders) | 10 | 0
Insomnia (Psychiatric disorders) | 13 | 2
Chromaturia (Renal and urinary disorders) | 3 | 3
Proteinuria (Renal and urinary disorders) | 7 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 10 | 4
Ovarian cyst (Reproductive system and breast disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 40 | 15
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Acne (Skin and subcutaneous tissue disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 3
Rash (Skin and subcutaneous tissue disorders) | 21 | 9
Rash papular (Skin and subcutaneous tissue disorders) | 7 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.